CLINICAL TRIAL: NCT03406260
Title: A Study to Investigate the Cardiovascular Effects of Lasmiditan in Healthy Elderly Subjects
Brief Title: A Study of Lasmiditan in Healthy Elderly Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17062; H8H-MC-LAIG (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-05

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lasmiditan 200 mg (milligrams) (Experimental): Participants received 200 mg of Lasmiditan tablet orally in the fasted state with approximately 240 (milliliter) mL of room temperature water in the morning of Days 1, 3, and 5, while participants were in a sitting position.
  Interventions: Drug: Lasmiditan
- Lasmiditan 100 mg (Experimental): Participants received 100 mg of Lasmiditan tablet orally in the fasted state with approximately 240 mL of room temperature water in the morning of Days 1, 3, and 5, while participants were in a sitting position.
  Interventions: Drug: Lasmiditan
- Placebo (Placebo Comparator): Participants received placebo tablet orally in the fasted state with approximately 240 mL of room temperature water in the morning of Days 1, 3, and 5, while participants were in a sitting position.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lasmiditan — Administered orally.
  Other Names: LY573144
  Arms: Lasmiditan 100 mg; Lasmiditan 200 mg (milligrams)
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The purposes of this study are to evaluate the effect of lasmiditan on blood pressure, as well as to look at the amount of study drug that gets into the blood stream and how long it takes the body to get rid of it in healthy elderly participants. The tolerability of the study drug will also be evaluated. Information about any side effects that may occur will also be collected. This study will take about 11 days, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined through medical history and physical examination
* Have a body mass index (BMI) of 19.0 to 35.0 kilograms per meter squared (kg/m²), inclusive, at the time of screening.

Exclusion Criteria:

* Have known allergies to lasmiditan, related compounds, or any components of the formulation.
* Are persons who have previously received lasmiditan.
* Have a history of, or electrocardiogram (ECG) findings of, clinically significant bradycardia, heart block, tachy or brady arrhythmias, or have any other abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data. appendectomy, splenectomy, and cholecystectomy are considered as acceptable.
* Show a history of central nervous system (CNS) conditions such as strokes, transient ischemic attacks, significant head trauma, seizures, CNS infections, migraines, brain surgery, or any other neurological conditions that, in the opinion of the investigator, increase the risk of participating in the study.
* Show evidence of active renal disease (e.g. diabetic renal disease, polycystic kidney disease) or estimated glomerular filtration rate <60 milliliters per minute per 1.73 meter squared (mL/min/m²).
* Have a history of syncope, presyncopy, uncontrolled vertigo, postural dizziness, or at risk for falls, as judged to be clinically significant by the investigator.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Covance Clinical Research Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover study with three study periods, each participant received single oral doses of Lasmiditan 200 milligrams (mg), Lasmiditan 100 mg and Placebo tablets as per the dosing sequence in each period. The washout period between dosing in consecutive study periods was at least 48 hours.
Groups:
- Sequence 1: Participants received Lasmiditan (200 milligrams (mg) and 100mg) and placebo tablets as per the below dosing schedule.
  Period 1: Lasmiditan 200 mg, Period 2: Lasmiditan 100 mg and Period 3: Placebo
- Sequence 2: Participants received Lasmiditan (200 milligrams (mg) and 100mg) and placebo tablets as per the below dosing schedule.
  Period 1: Lasmiditan 100 mg, Period 2: Placebo and Period 3: Lasmiditan 200 mg
- Sequence 3: Participants received Lasmiditan (200 milligrams (mg) and 100mg) and placebo tablets as per the below dosing schedule.
  Period 1: Placebo, Period 2: Lasmiditan 200 mg and Period 3: Lasmiditan 100 mg
- Sequence 4: Participants received Lasmiditan (200 milligrams (mg) and 100mg) and placebo tablets as per the below dosing schedule.
  Period 1: Placebo, Period 2: Lasmiditan 100 mg and Period 3: Lasmiditan 200 mg
- Sequence 5: Participants received Lasmiditan (200 milligrams (mg) and 100mg) and placebo tablets as per the below dosing schedule.
  Period 1: Lasmiditan 200 mg, Period 2: Placebo and Period 3: Lasmiditan 100 mg
- Sequence 6: Participants received Lasmiditan (200 milligrams (mg) and 100mg) and placebo tablets as per the below dosing schedule.
  Period 1: Lasmiditan 100 mg, Period 2: Lasmiditan 200 mg and Period 3: Placebo
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 6 | 6 | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 6 | 6 | 6 | 5 | 6
Completed | 6 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 6 | 6 | 6 | 5 | 6
Completed | 6 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 0 | 0 | 0 | 2
  >=65 years | 5 | 5 | 6 | 6 | 6 | 6 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 2 | 4 | 15
  Male | 4 | 4 | 4 | 3 | 4 | 2 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 6 | 5 | 6 | 5 | 5 | 6 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1 | 2
  White | 5 | 6 | 6 | 6 | 6 | 5 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics: Change From Baseline in Peak Hourly Mean Values of Systolic Blood Pressure (SBP)
Description: Mean 24-hour systolic blood pressure (SBP) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Ambulatory blood pressure measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using linear mixed effects model adjusting for baseline, treatment, treatment sequence, period, treatment by time point interaction, and a random effect of participant.
Time Frame: Baseline through 24 hours after each administration of study drug
Population: All randomized participants who received at least one dose of study drug and have data for SBP
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Groups:
- Lasmiditan 200 mg: Participants received 200 mg of Lasmiditan tablet orally in the fasted state with approximately 240 (milliliters) mL of room temperature water in the morning of Days 1, 3, and 5, while participants were in a sitting position.
Arm/Group | Lasmiditan 200 mg | Lasmiditan 100 mg | Placebo
Number analyzed (Participants) | 36 | 34 | 35
millimeters of mercury (mmHg) | 15.79 (1.774) | 15.50 (1.820) | 17.14 (1.797)
Statistical Analysis 1: Comparison: Lasmiditan 100 mg vs Placebo; Test type: Non-Inferiority — A p-value < 0.05 indicates lasmiditan can be declared noninferior to placebo with noninferiority margin of 10 mmHg, i.e. the difference lasmiditan mean minus placebo mean is less than 10 mmHg; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference (Final Vaules) = -1.63, 95% CI 2-sided [-1000 to 1.81]
Statistical Analysis 2: Comparison: Lasmiditan 200 mg vs Placebo; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference (Final Vaules) = -1.35, 95% CI 2-sided [-1000 to 2.06]

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Lasmiditan
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Lasmiditan.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours, postdose
Population: All randomized participants who received at least one dose of study drug and have evaluable pharmacokinetics (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Lasmiditan 200 mg: Participants received 200 mg of Lasmiditan tablet orally in the fasted state with approximately 240 mL of room temperature water in the morning of Days 1, 3, and 5, while participants were in a sitting position.
Arm/Group | Lasmiditan 100 mg | Lasmiditan 200 mg
Number analyzed (Participants) | 35 | 36
nanogram per milliliter (ng/mL) | 159 (32) | 339 (34)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Lasmiditan
Description: PK: Area under the Concentration Versus Time Curve from Zero to Infinity (AUC[0-∞]) of Lasmiditan.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours, postdose
Population: All randomized participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Lasmiditan 100 mg | Lasmiditan 200 mg
Number analyzed (Participants) | 35 | 36
nanogram*hour per milliliter (ng*h/mL) | 1170 (34) | 2470 (35)

ADVERSE EVENTS:
Time Frame: Up To 12 days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Lasmiditan 200 mg | Lasmiditan 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 15/36 | 6/35 | 0/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lasmiditan 200 mg (N=36) | Lasmiditan 100 mg (N=35) | Placebo (N=35)
Fatigue (General disorders) | 4 (4) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 9 (9) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the Study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.

DOCUMENTS (2):
  • Study Protocol (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03406260/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT03406260/SAP_001.pdf